CLINICAL TRIAL: NCT03257124
Title: An Open Label, Multicenter, Phase II Study of AZD9291 in Non-small Cell Lung Cancer (NSCLC) Patients Harboring T790M Mutation Who Failed EGFR TKIs and With Brain and/or Leptomeningeal Metastasis
Brief Title: Study of AZD9291 in NSCLC Patients Harboring T790M Mutation Who Failed EGFR TKI and With Brain and/or LMS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Myung-Ju Ahn, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-09-058
Record Dates: First submitted 2017-05-07; First posted 2017-08-22 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Non-Small Cell Lung Cancer With EGFR T790M Mutation; With Brain and/or Leptomeningeal Metastasis; Failed Tyrosine Kinase Inhibitors
MeSH Terms: interventions — osimertinib

STUDY DESIGN:
Intervention Model Description: 1. Brain Metastasis cohort (BM cohort)
  2. Leptomeningeal Metastasis cohort (LM cohort)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AZD9291 in BM or LM cohort in T790M positive (Experimental): 1. Brain metastasis cohort (BM cohort)
  2. Leptomeningeal metastasis cohort (LM cohort)
  Interventions: Drug: AZD9291

INTERVENTIONS:
Drug: AZD9291 — AZD9291 160mg per oral daily (1 cycle of 28 days)
  Other Names: Osimertinib

SUMMARY:
AZD9291 is an oral potent irreversible EGFR TKI selective for sensitizing EGFR mutation and T790M resistance mutation but sparing wild-type EGFR. Preclinical studies indicate that AZD9291 has significant exposure in the brain and activity against EGFR mutant brain metastasis. In addition, anti-tumor activities of AZD9291 in patients with advanced stage EGFR mutant NSCLC including patients with brain metastasis have been reported in an ongoing Phase I study. More recently, AZD9291 at a dose of 160mg also showed promising efficacy in heavily pre-treated patients with leptomeningeal disease from EGFR mutant NSCLC. Among 11 evaluable for response, 6 patients had LM imaging improvement and 3 out of 7 patients with abnormal neurological exam at baseline had symptomatic improvement. Compared to AZD9291, other 3rd generation EGFR TKIs, rociletinib or HM61713 has not been reported to be effective in most of CNS disease of NSCLC. Further, previous studies with AZD9291 showed anecdotal case series or undetermined for T790M mutation status, indicating more systematic study is warranted.

Based on these data, the investigators are going to conduct phase II study of AZD9291 in NSCLC patients harboring T790M mutation who failed EGFR TKIs and brain and/or leptomeningeal metastasis.

DETAILED DESCRIPTION:
1. Primary end points

   * Overall response rate (ORR) in CNS -brain metastasis cohort
   * Overall survival - Leptomeningeal with or without brain metastasis cohort
2. Secondary end points

   * Whole body disease control rate (DCR)
   * Time to brain progression
   * Progression free survival (PFS) in BM cohort
   * Overall survival (OS)
   * Adverse events (AEs)
   * Exploratory analysis of EGFR mutation/T790M in tissue, plasma or cerebrospinal fluid (CSF)
3. Treatment AZD9291 160mg po daily (1 cycle of 28 days)
4. Total patient sample size Eligible patients will be divided into two cohorts, brain metastasis (BM) cohort and leptomeningeal metastasis (LM) with or without BM cohort. The two patient cohorts use different primary endpoints.
5. BM cohort For the BM cohort, the primary outcome is overall response (CR+PR). Let P denote the overall response rate of AZD9291. From some preliminary data of response in the brain or leptomeningeal seeding with AZD 9291 in phase II AURA and BLOOM study, we hypothesized that H0:P= 10% and H1:P =30%. The BM cohort uses Simon's optimal two-stage design as follows.

   Stage 1: Treat n1 = 18 patients. If r1 = 2 or fewer patients respond, stop the BM cohort concluding that the study therapy is inefficacious. Otherwise, proceed to Stage 2.

   Stage 2: Treat additional n2 = 17 patients. If r = 6 or fewer patients respond among the cumulative n1 + n2 = 35 patients, then conclude that the study therapy is inefficacious. Otherwise, accept the study therapy for further investigation.

   This design has 1-sided alpha = 5% for P0 = 10% and power = 90% for P1 = 30%. Considering about 10%, of attrition due to ineligibility and dropout, a total of 40 patients will be enrolled into the BM cohort.
6. LM ± BM cohort

   The primary outcome of the LM ± BM cohort is overall survival (OS). Let μ denote the median OS of AZD9291 in this cohort. Based on some preliminary results (we need a reference), we hypothesize that H0: μ=3 months vs. H1: μ=5 months. Assuming an exponential OS distribution under H0, the investigators will conduct the 1-sample log-rank test. In this cohort, the investigators expect an accrual rate of 30 patients per year and about 10% of attrition, and will have an additional follow-up of 6 months after completion of accrual. Under these assumptions, we need N=40 patients (D=29 deaths) for 90% of power by the 1-sample log-rank test with 1-sided alpha=5% (refer to Kwak and Jung 2013). The trial of this cohort is expected to take about 22 months (=16 months for patient accrual + 6 months for additional follow-up).
7. Statistical analysis plan

The analysis is conducted separately for each cohort. OS, PFS, and time to brain progression will be summarized by Kaplan-Meier method. DCR and AEs will be summarized using contingency tables. Cohort specific analyses are conducted as follows.

BM cohort

Two-stage testing on ORR will be conducted as described in "Target number" section. If the final sample size is different from n1=18 or n1 + n2=35, then a 1-sided p-value will be calculated by Jung et al. (2006) and accept the experimental therapy if it is smaller than alpha = 5%. The ORR will be unbiasedly estimated by Jung and Kim (2004), and its confidence interval will be calculated by Jennison and Turnbull (1983).

LM ± BM cohort

The final analysis of this cohort will be conducted when D29 deaths are observed, which is expected to be about 22 months from the study open. The investigators will conduct a 1-sample log-rank test assuming the exponential OS distribution with a median of 3 months under H0.

ELIGIBILITY:
Inclusion Criteria:

* EGFR activating mutant NSCLC patients who failed EGFR TKIs (gefitinib, erlotinib, or afatinib) and develop CNS disease (BM and/or LM) with T790M mutation either tissue or plasma. For patients with intracranial progression, prior radiation therapy is not mandatory. Extracranial progression is allowed.
* Patients who failed to 3rd generation EGFR TKIs (AZD9291 (80mg), Rociletinib, HM61713) and develop CNS progression but stable extracranial disease
* Age ≥18 years
* ECOG performance status of 0 to 2
* For BM, at least one measurable intracranial lesion as ≥ 10mm in the longest diameter by magnetic resonance imaging (MRI)
* For LM, at least one site of CNS leptomeningeal disease that can be assessed by MRI
* Adequate organ function as evidenced by the following;

  * Absolute neutrophil count > 1.5 x 109/L;
  * platelets > 100 x 109/L;
  * total bilirubin ≤1.5 UNL;
  * AST and/or ALT < 5 UNL;
  * CCr ≥ 50mL/min.
* Female subjects must either be of non-reproductive potential
* Subject is willing and able to comply with the protocol
* Signed written informed consent

Exclusion Criteria:

* Radiotherapy with a wide field of radiation within 4 weeks or radiotherapy with a limited field of radiation for palliation within 1 week
* Any unresolved toxicities from prior therapy, greater than CTCAE grade 1
* Mean QT interval corrected for heart rate (QTc) ≥ 470 ms
* Uncontrolled systemic illness including uncontrolled hypertension, active bleeding, or active infection.
* Past medical history of interstitial lung disease, drug induced interstitial lung disease, radiation pneumonitis which required steroid treatment
* History of hypersensitivity to AZD9291
* Known intracranial haemorrahge which is unrelated to tumor Refractory nausea and vomiting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) in CNS -brain metastasis cohort | December, 2019 (one-year follow-up from last patient -in)
  At least one visit response of CR (complete response) or PR (partial response) that is confirmed at least 4 weeks later by using RECIST 1.1 criteria
Overall survival - Leptomeningeal with or without brain metastasis cohort | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  From the date of study start to the date of all cause death

SECONDARY OUTCOMES:
Whole body disease control rate (DCR) | December, 2019 (one-year follow-up from last patient -in)
  At least one visit response of CR (complete response), PR (partial response) or SD (stable disease) that is confirmed at least 4 weeks later by using RECIST 1.1 criteria.
Time to brain progression | December, 2019 (one-year follow-up from last patient -in)
  Time to brain progression is measured from the date of start of study to the date of progression of BM or LM.
Progression free survival (PFS) in BM cohort | December, 2019 (one-year follow-up from last patient -in)
  measured from the date of start of study to the date of disease progression or death from any cause.
Overall survival (OS) | December, 2019 (one-year follow-up from last patient -in)
  OS is measured from the date of start of study to the date of death from any cause
Adverse events (AEs) | December, 2019 (one-year follow-up from last patient -in)
  Adverse events will be measured by the CTCAE scale, version 4.
Exploratory analysis of EGFR mutation/T790M | December, 2019 (one-year follow-up from last patient -in)
  Exploratory analysis of EGFR mutation/T790M in tissue, plasma or cerebrospinal fluid (CSF)

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Ju Ahn, Professor, Principal Investigator — Samsung Medical Center
Locations (1):
- Department of Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mok TS, Wu YL, Thongprasert S, Yang CH, Chu DT, Saijo N, Sunpaweravong P, Han B, Margono B, Ichinose Y, Nishiwaki Y, Ohe Y, Yang JJ, Chewaskulyong B, Jiang H, Duffield EL, Watkins CL, Armour AA, Fukuoka M. Gefitinib or carboplatin-paclitaxel in pulmonary adenocarcinoma. N Engl J Med. 2009 Sep 3;361(10):947-57. doi: 10.1056/NEJMoa0810699. Epub 2009 Aug 19. PMID 19692680
- [Background] Bonomi PD. Implications of key trials in advanced nonsmall cell lung cancer. Cancer. 2010 Mar 1;116(5):1155-64. doi: 10.1002/cncr.24815. PMID 20087963
- [Background] Mok TS. Personalized medicine in lung cancer: what we need to know. Nat Rev Clin Oncol. 2011 Aug 23;8(11):661-8. doi: 10.1038/nrclinonc.2011.126. PMID 21862980
- [Background] Lee SJ, Lee JI, Nam DH, Ahn YC, Han JH, Sun JM, Ahn JS, Park K, Ahn MJ. Leptomeningeal carcinomatosis in non-small-cell lung cancer patients: impact on survival and correlated prognostic factors. J Thorac Oncol. 2013 Feb;8(2):185-91. doi: 10.1097/JTO.0b013e3182773f21. PMID 23328548
- [Background] Lee E, Keam B, Kim DW, Kim TM, Lee SH, Chung DH, Heo DS. Erlotinib versus gefitinib for control of leptomeningeal carcinomatosis in non-small-cell lung cancer. J Thorac Oncol. 2013 Aug;8(8):1069-74. doi: 10.1097/JTO.0b013e318294c8e8. PMID 23804027
- [Background] Gow CH, Chien CR, Chang YL, Chiu YH, Kuo SH, Shih JY, Chang YC, Yu CJ, Yang CH, Yang PC. Radiotherapy in lung adenocarcinoma with brain metastases: effects of activating epidermal growth factor receptor mutations on clinical response. Clin Cancer Res. 2008 Jan 1;14(1):162-8. doi: 10.1158/1078-0432.CCR-07-1468. PMID 18172267
- [Background] Wu YL, Zhou C, Cheng Y, Lu S, Chen GY, Huang C, Huang YS, Yan HH, Ren S, Liu Y, Yang JJ. Erlotinib as second-line treatment in patients with advanced non-small-cell lung cancer and asymptomatic brain metastases: a phase II study (CTONG-0803). Ann Oncol. 2013 Apr;24(4):993-9. doi: 10.1093/annonc/mds529. Epub 2012 Nov 4. PMID 23129122
- [Background] Umemura S, Tsubouchi K, Yoshioka H, Hotta K, Takigawa N, Fujiwara K, Horita N, Segawa Y, Hamada N, Takata I, Yamane H, Kamei H, Kiura K, Tanimoto M. Clinical outcome in patients with leptomeningeal metastasis from non-small cell lung cancer: Okayama Lung Cancer Study Group. Lung Cancer. 2012 Jul;77(1):134-9. doi: 10.1016/j.lungcan.2012.03.002. Epub 2012 Apr 7. PMID 22487432
- [Background] Pao W, Miller VA, Politi KA, Riely GJ, Somwar R, Zakowski MF, Kris MG, Varmus H. Acquired resistance of lung adenocarcinomas to gefitinib or erlotinib is associated with a second mutation in the EGFR kinase domain. PLoS Med. 2005 Mar;2(3):e73. doi: 10.1371/journal.pmed.0020073. Epub 2005 Feb 22. PMID 15737014
- [Background] Planchard D, Loriot Y, Andre F, Gobert A, Auger N, Lacroix L, Soria JC. EGFR-independent mechanisms of acquired resistance to AZD9291 in EGFR T790M-positive NSCLC patients. Ann Oncol. 2015 Oct;26(10):2073-8. doi: 10.1093/annonc/mdv319. Epub 2015 Aug 12. PMID 26269204
- [Background] Janne PA, Yang JC, Kim DW, Planchard D, Ohe Y, Ramalingam SS, Ahn MJ, Kim SW, Su WC, Horn L, Haggstrom D, Felip E, Kim JH, Frewer P, Cantarini M, Brown KH, Dickinson PA, Ghiorghiu S, Ranson M. AZD9291 in EGFR inhibitor-resistant non-small-cell lung cancer. N Engl J Med. 2015 Apr 30;372(18):1689-99. doi: 10.1056/NEJMoa1411817. PMID 25923549
- [Background] Cross DA, Ashton SE, Ghiorghiu S, Eberlein C, Nebhan CA, Spitzler PJ, Orme JP, Finlay MR, Ward RA, Mellor MJ, Hughes G, Rahi A, Jacobs VN, Red Brewer M, Ichihara E, Sun J, Jin H, Ballard P, Al-Kadhimi K, Rowlinson R, Klinowska T, Richmond GH, Cantarini M, Kim DW, Ranson MR, Pao W. AZD9291, an irreversible EGFR TKI, overcomes T790M-mediated resistance to EGFR inhibitors in lung cancer. Cancer Discov. 2014 Sep;4(9):1046-61. doi: 10.1158/2159-8290.CD-14-0337. Epub 2014 Jun 3. PMID 24893891
- [Derived] Park S, Lee MH, Seong M, Kim ST, Kang JH, Cho BC, Lee KH, Cho EK, Sun JM, Lee SH, Ahn JS, Park K, Ahn MJ. A phase II, multicenter, two cohort study of 160 mg osimertinib in EGFR T790M-positive non-small-cell lung cancer patients with brain metastases or leptomeningeal disease who progressed on prior EGFR TKI therapy. Ann Oncol. 2020 Oct;31(10):1397-1404. doi: 10.1016/j.annonc.2020.06.017. Epub 2020 Jul 5. PMID 32634610